CLINICAL TRIAL: NCT06831851
Title: The Influence of Music and Storytelling on the Linguistic, Socioemotional, and Adaptive Development of Children Aged 12-36 Months: an Intervention Protocol in an Enriched Environment Conducted in Municipal Early Childhood Education Centers (CMEIs)
Brief Title: Effects of Music and Storytelling on Linguistic, Socioemotional, and Adaptive Development in Children Aged 12-36 Months: an Intervention Protocol in Municipal Early Childhood Centers
Acronym: MUS-STORY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Aline A de Lima, MA, Principal Investigator, MSc in Neuroscience, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INF-MUSIC-STORY01
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Child Development; Adaptive Behavior; Early Child Development; Music Education; Preschool Education
Keywords: Environmental enrichment; Child development; Early childhood education; Adaptive behavior; Randomized clinical trial

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: No other parties are masked in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group with Parental Guidance (Experimental): Children in this group will participate in structured storytelling sessions (30 minutes per day, once a week) and music education activities (40 minutes, twice per week) in an enriched learning environment. The intervention aims to enhance cognitive, linguistic, socio-emotional, and motor development.
  Additionally, parents or guardians will attend 8 biweekly guidance sessions (60 minutes each), where they will be trained in strategies to reinforce storytelling and musical activities at home. These sessions will provide tools to improve parent-child interaction and promote continuity of learning beyond the daycare setting
  Interventions: Behavioral: Storytelling Sessions; Behavioral: Music Education Sessions; Behavioral: Parental Guidance Sessions
- Intervention Group without Parental Guidance (Experimental): Children in this group will participate in structured storytelling sessions (30 minutes per day, once a week) and music education activities (40 minutes, twice per week) in an enriched learning environment. The intervention is designed to stimulate cognitive, linguistic, socio-emotional, and motor development through interactive and engaging activities.
  Unlike the parental guidance group, this intervention does not include parental training sessions. The activities will be conducted exclusively in the daycare setting, without reinforcement at home
  Interventions: Behavioral: Storytelling Sessions; Behavioral: Music Education Sessions
- Control Group (Active Comparator): Children in this group will receive standard daycare activities without structured intervention. Activities will include artistic and pedagogical tasks (e.g., drawing, painting, modeling) as part of their regular curriculum. Additionally, storytelling will be conducted once a week, but without a structured approach or the integration of music education as applied in the experimental groups.
  This group serves as a comparator to assess the effects of storytelling and music education interventions on cognitive, linguistic, socio-emotional, and motor development
  Interventions: Behavioral: Standard Daycare Activities

INTERVENTIONS:
Behavioral: Storytelling Sessions — Children will participate in structured storytelling sessions, held once a week for 30 minutes per session. The sessions will use interactive narrative techniques, including voice modulation, gestures, and visual aids, to enhance cognitive, linguistic, and socio-emotional development. The intervention is designed to promote active engagement, stimulate imagination, and improve attention and language skills in early childhood.
  Arms: Intervention Group with Parental Guidance; Intervention Group without Parental Guidance
Behavioral: Music Education Sessions — Children will participate in structured music education sessions, conducted twice per week for 40 minutes each. The sessions will include rhythm exercises, vocalization, body percussion, and instrumental exploration using age-appropriate musical instruments. Activities will be designed to enhance cognitive, motor, and socio-emotional development by fostering auditory discrimination, fine and gross motor coordination, and social interaction. The intervention follows an interactive and play-based methodology, ensuring active engagement and progressive learning.
  Arms: Intervention Group with Parental Guidance; Intervention Group without Parental Guidance
Behavioral: Parental Guidance Sessions — Parents or guardians will attend 8 biweekly training sessions (60 minutes each) designed to equip them with strategies for cognitive, linguistic, and socio-emotional stimulation in early childhood. The sessions will include practical guidance on storytelling techniques, musical interaction, and play-based learning to reinforce the intervention at home. The goal is to create continuity between structured intervention activities and the home environment, maximizing developmental outcomes for the children. Sessions will be interactive, combining theoretical content with practical exercises and demonstrations
  Arms: Intervention Group with Parental Guidance
Behavioral: Standard Daycare Activities — Children in this group will participate in regular daycare activities, including artistic and pedagogical tasks such as drawing, painting, and modeling. These activities are part of the standard curriculum and do not include structured storytelling or music education interventions
  Arms: Control Group

SUMMARY:
This randomized clinical trial aims to evaluate the impact of a structured enriched environment on the linguistic, adaptive behavior, and socioemotional development of children aged 12 to 36 months. The study addresses two main questions:

Does the intervention improve linguistic, adaptive behavior, and socioemotional development compared to standard care? Does parental guidance amplify the benefits of the intervention?

Participants will be randomly assigned to one of two groups:

Intervention Group:

Children will participate in musical activities twice per week (singing, exploring simple instruments, and musical games) and daily storytelling sessions using interactive and visual aids.

Within this group, parents in the "with guidance" subgroup will attend biweekly meetings to learn strategies for reinforcing the intervention at home, while the "without guidance" subgroup will not include parental training.

Control Group:

Children will receive standard care complemented by alternative artistic and pedagogical activities (e.g., drawing, painting), without the structured intervention.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of an enriched intervention program on early childhood development, emphasizing the role of parental involvement. Participants will be randomly assigned to two main groups:

Control Group:

Children will follow routine childcare activities, including artistic and educational engagements (e.g., drawing, painting, storytelling).

Intervention Group:

Children in this group will participate in a structured program combining daily storytelling sessions and weekly musicalization activities.

This group will be further divided into two subgroups:

With Parental Guidance: Parents or guardians will attend bi-weekly guidance meetings to receive strategies for reinforcing the intervention at home.

Without Parental Guidance: No parental meetings will be conducted; children will participate in the program independently.

Intervention Activities:

The intervention includes:

Storytelling: Interactive, daily sessions (30 minutes/day) designed to foster creativity and imagination using visual and verbal methods.

Musicalization: Interactive, twice-weekly sessions (40 minutes each) incorporating singing, rhythm games, and exploration of simple musical instruments to enhance motor and cognitive skills.

Assessment Measures:

The primary developmental domains-linguistic, socio-emotional, and adaptive behaviors-will be assessed using the Bayley Scales of Infant and Toddler Development (Bayley-III). Secondary measures include parental adherence (in the guidance subgroup) and engagement levels during activities.

This pilot study will provide foundational data to support the development of larger-scale, evidence-based interventions focused on enhancing early childhood developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

Children of both sexes, aged between 12 and 36 months. Enrolled full-time in Municipal Early Childhood Education Centers (CMEIs). Attending with a daily workload of 10 hours, five days a week.

Exclusion Criteria:

Diagnosis of atypical neurodevelopment. Use of sedative or stimulant medications for memory. Undergoing physical therapy for the locomotor system. Presence of any clinical or functional condition that prevents participation. More than five consecutive absences from the intervention program.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Developmental Assessment using Bayley-III Scales of Infant and Toddler Development | The primary outcome measure (developmental assessment using Bayley-III) will be assessed at baseline (before the intervention) and after 4 months of intervention, focusing on linguistic, socio-emotional, and adaptive behavior domains
  Developmental Assessment using the Bayley-III Scales The primary outcome measure will focus on evaluating the child's development through the Bayley Scales of Infant and Toddler Development (Bayley-III), a widely used tool for assessing multiple domains of early childhood development, including cognitive, motor, language, socio-emotional, and adaptive behavior. The aim is to detect any developmental delays or deviations, providing critical information for early intervention. The Bayley-III will be administered to children up to 42 months of age to ensure comprehensive developmental screening across different stages.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco (UFPE) - Department of Neuropsychiatry and Behavioral Sciences, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR